CLINICAL TRIAL: NCT01234363
Title: Evaluation of the Potential of Elastography for Noninvasive Assessment of Fibrosis in Kidney Transplant
Brief Title: Renal Allograft : Evaluation of Parenchymal Fibrosis by Elastography
Acronym: GREFE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009.590
Record Dates: First submitted 2010-07-26; First posted 2010-11-04 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Renal Transplant
Keywords: Renal allograft; kidney; fibrosis; elastography; elasticity
MeSH Terms: conditions — Fibrosis | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Magnetic Resonance Elastography, Supersonic Shear Imaging (Experimental): Magnetic Resonance Elastography and Supersonic Shear Imaging
  Interventions: Device: Magnetic Resonance Elastography, and Supersonic Shear Imaging

INTERVENTIONS:
Device: Magnetic Resonance Elastography, and Supersonic Shear Imaging — Magnetic Resonance Elastography, and Supersonic Shear Imaging

SUMMARY:
The purpose of this study is to assess the potential of elastography for noninvasive assessment of fibrosis in renal allograft.

ELIGIBILITY:
Inclusion Criteria:

* Renal allograft performed less than 3 months before enrolment

Exclusion Criteria:

* Contra-indication to magnetic resonance imaging
* Contra-indication to biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-05; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Correlation between elasticity (as measured by elastography) and (a) Banff score for fibrosis, (b) glomerular filtration rate assessed by creatinine clearance, (c) glomerular filtration rate assessed by insulin clearance | 3 months and 12 months after graft

SECONDARY OUTCOMES:
Number of technical failures | 12 months
Tolerance (assessed by a questionnaire) | 3 months and 12 months after graft
Evolution of the elasticity of the transplant between 3 and 12 months after graft | 3 months and 12 months after graft
Correlation between elasticity and arterial resistance index | 3 months and 12 months after graft

CONTACTS AND LOCATIONS:
Overall Officials: ROUVIERE Olivier, Pr, Principal Investigator — Hospices Civils de Lyon Service de Radiologie, Pavillon P Radio, Hôpital Edouard Herriot, 69437 Lyon Cedex 03
Locations (1):
- Service de Radiologie, Pavillon P Radio, Hôpital Edouard Herriot, Lyon, Lyon, France